CLINICAL TRIAL: NCT03453502
Title: Improving Mother Milk Feeding Benefits in Neonatal Intensive Care Units Using the Evidence-based Practice for Quality Improvement
Brief Title: Improving Mother Milk Feeding Benefits in Neonatal Intensive Care Units
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: Nanjing Maternity and Child Health Care Hospital (Other); Jiangsu Women and Children Health Hospital (Unknown); The First People's Hospital of Lianyungang (Other); Xuzhou Maternity and Child Health Care Hospital (Other); The Second Hospital of Nanjing Medical University (Other); Children's Hospital of Nanjing Medical University (Other); Suqian Maternity and Child Health Care Hospital (Unknown); Lianyungang Maternity and Child Health Care Hospital (Unknown); Wuxi Women's & Children's Hospital (Other); Suzhou Municipal Hospital (Other); Yancheng Maternity and Child Health Care Hospital (Unknown); The First People's Hospital of Yancheng (Unknown); The Affiliated Jiangyin Hospital of Southeast University Medical College (Unknown); The First People's Hospital of Zhangjiagang (Unknown); The Affiliated Huaian NO.1 People's Hospital of Nanjing Medical University (Unknown); Huaian Maternity and Child Health Care Hospital (Unknown); Changzhou Maternal and Child Care Hospital (Other); Zhenjiang Maternity and Child Health Care Hospital (Unknown); The Affiliated Hospital of Xuzhou Medical University (Other); Taizhou People's Hospital (Unknown); Affiliated Hospital of Jiangsu University (Other); First People's Hospital of Hangzhou (Other); Wuxi Maternity and Child Health Care Hospital (Unknown); Changzhou Children's Hospital (Unknown); Northern Jiangsu People's Hospital (Other); Children's Hospital of Soochow University (Other); Nantong Maternity and Child Health Care Hospital (Unknown)
Responsible Party: Principal Investigator, Zhangbin Yu, Principal Investigator, Nanjing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NMU-FY2017-350
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Quality Improvement; Breast Milk
Keywords: quality improvement; breast milk

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Before-intervention phase (No Intervention): All the very low birth weight (VLBW) and extremely low birth weight (ELBW) infants who were admitted from January 2017 to December 2017 to the NICUs of different hospitals.
- Intervention phase (Experimental): All the VLBW and ELBW infants who were admitted from January 2018 to December 2018 to the NICUs.During this phase,multiple intervention bundles of quality improvement will be implemented.
  Interventions: Behavioral: Quality improvement of breast milk feeding
- Sustainability intervention phase (Experimental): All the VLBW and ELBW infants who were admitted from January 2019 to December 2019to the NICUs.In the Sustainability intervention phase,multiple intervention bundles of quality improvement will be continuous implemented.
  Interventions: Behavioral: Quality improvement of breast milk feeding

INTERVENTIONS:
Behavioral: Quality improvement of breast milk feeding — During the Intervention phase and Sustainability phase ,The NICUs will receive training of multiple evidence based quality improvement methods.
  Arms: Intervention phase; Sustainability intervention phase

SUMMARY:
Twenty-seven hospitals in China will participate in the study, which aims to increase breastfeeding rate in the neonatal intensive care unit (NICU) and reduce the clinical complications in very low birth weight infants and extremely low birth weight infants.

DETAILED DESCRIPTION:
Breast milk reduces the risk of serious prematurity related morbidities. Quality improvement is an effective means of increasing breast milk feeding.Twenty-seven hospitals in China will participate in the study, which aims to increase breastfeeding rate in the NICU and reduce the clinical complications in very low birth weight infants and extremely low birth weight infants. This study compared the clinical data of very low birth weight infants and extremely low birth weight infants in three phases：Before-intervention phase，Intervention phase and Sustainability phase. During the Intervention phase and Sustainability phase multiple intervention bundles of quality improvement were implemented.The investigators will compare breast milk feeding rate and neonatal outcomes in different phases.

ELIGIBILITY:
Inclusion Criteria:

* premature Infants (Birth weight<1500g)

Exclusion Criteria:

* mother with sever illness or communicable disease

Max Age: 120 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1800 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
mother own milk feeding rates | three years

SECONDARY OUTCOMES:
NICU costs | three years
  costs during hospitalization in NICU
the incidence of necrotizing enterocolitis (NEC) | three years
  the incidence of necrotizing enterocolitis
the incidence of sepsis | three years
Reduce the incidence of enteral feed intolerance | three years

CONTACTS AND LOCATIONS:
Overall Officials: Shuping Han, PhD, Study Director — Nanjing Maternity and Child Health Care Hospital; Zhangbin Yu, PhD, Study Director — Nanjing Maternity and Child Health Care Hospital; Jun Zhang, PhD, Principal Investigator — Nanjing Maternity and Child Health Care Hospital; Yuhua Hu, PhD, Principal Investigator — Jiangsu Women and Children Health Hospital; Shan Li, PhD, Principal Investigator — The First People's Hospital of Lianyungang; Xiaoyi Deng, PhD, Principal Investigator — Xuzhou Maternity and Child Health Care Hospital; Zelin Jiao, PhD, Principal Investigator — The Second Hospital of Nanjing Medical University; Rui Cheng, PhD, Principal Investigator — Children's Hospital of Nanjing Medical University; Weiyuan Wang, PhD, Principal Investigator — Suqian Maternity and Child Health Care Hospital; Yan Gao, PhD, Principal Investigator — Lianyungang Maternity and Child Health Care Hospital; Zhengying Li, PhD, Principal Investigator — Wuxi Women's & Children's Hospital; Sannan Wang, PhD, Principal Investigator — Suzhou Municipal Hospital; Jinlan Chai, PhD, Principal Investigator — Yancheng Maternity and Child Health Care Hospital; Zhun xu, PhD, Principal Investigator — The First People's Hospital of Yancheng; Jun Wan, PhD, Principal Investigator — The Affiliated Jiangyin Hospital of Southeast University Medical College; Weidong xu, PhD, Principal Investigator — The First People's Hospital of Zhangjiagang; Zhaofang Tian, PhD, Principal Investigator — The Affiliated Huaian NO.1 People's Hospital of Nanjing Medical University; Liangrong Han, PhD, Principal Investigator — Huaian Maternity and Child Health Care Hospital; Jinxiu Wang, PhD, Principal Investigator — Changzhou Maternal and Child Care Hospital; Xuqin Mao, PhD, Principal Investigator — Zhenjiang Maternity and Child Health Care Hospital; Jun Wang, PhD, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University; Mei Xue, PhD, Principal Investigator — Taizhou People's Hospital; Hongyan Lu, PhD, Principal Investigator — Affiliated Hospital of Jiangsu University; Mingfu Wu, PhD, Principal Investigator — First People's Hospital of Hangzhou; Qin Zhou, PhD, Principal Investigator — Wuxi Maternity and Child Health Care Hospital; Wenjuan Tu, PhD, Principal Investigator — Changzhou Children's Hospital; Lingling Zhu, PhD, Principal Investigator — Northern Jiangsu People's Hospital; Bin Sun, PhD, Principal Investigator — Children's Hospital of Soochow University; Shuangshuang Li, PhD, Principal Investigator — Nantong Maternity and Child Health Care Hospital; Xiaohui Chen, PhD, Principal Investigator — Nanjing Maternity and Child Health Care Hospital

REFERENCES:
- [Derived] Xu Y, Yu Z, Li Q, Zhou J, Yin X, Ma Y, Yin Y, Jiang S, Zhu R, Wu Y, Han L, Gao Y, Xue M, Qiao Y, Zhu L, Tu W, Wu M, Wan J, Wang W, Deng X, Li S, Wang S, Chen X, Zhou Q, Wang J, Cheng R, Wang J, Han S. Dose-dependent effect of human milk on Bronchopulmonary dysplasia in very low birth weight infants. BMC Pediatr. 2020 Nov 16;20(1):522. doi: 10.1186/s12887-020-02394-1. PMID 33190629